CLINICAL TRIAL: NCT05278364
Title: A Phase I/II, Open-Label, Single-arm, Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antineoplastic Activity of SY-5007 in Patients With RET-altered Advanced Solid Tumor.
Brief Title: Phase I/II Study of SY-5007, a RET Inhibitor, in Patients With RET-altered Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SY-5007-I
Record Dates: First submitted 2022-03-08; First posted 2022-03-14 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Non-Small Cell Lung Cancer; Medullary Thyroid Cancer; Solid Tumor
Keywords: SY-5007; RET-fusion positive NSCLC; RET-mutant MTC; RET-altered advanced solid tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Medullary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-escalation and Dose-expansion (Experimental): Dose-escalation Phase:
  Multiple doses of SY-5007 for oral administration.
  Dose Expansion Phase:
  RP2D of SY-5007 as determined during Dose Escalation.
  Interventions: Drug: SY-5007

INTERVENTIONS:
Drug: SY-5007 — a RET selective Inhibitor
  Other Names: SY-5007 Capsule

SUMMARY:
This is a phase I/II, open-label, multi-center, first-in-human study designed to evaluate the safety, tolerability, pharmacokinetics (PK) and preliminary anti-tumor activity of SY-5007 administered orally to participants with advanced solid tumors, including RET Fusion-Positive NSCLC or RET-mutated MTC or other RET-altered advanced solid tumor.

DETAILED DESCRIPTION:
The study consists of 2 parts:

Part 1: Dose-escalation and dose-expansion in patients with RET Fusion-Positive NSCLC or RET-mutated MTC or other RET-altered advanced solid tumor. Dose-escalation study phase is designed to determine the DLTs (Dose-limiting toxicity) and recommended phase II dose (RP2D) and to characterize the safety, tolerability, and pharmacokinetics (PK) profile of SY-5007. Dose-expansion study phase is designed to evaluate the antitumor activity (ORR, DCR and DoR) of SY-5007 in patients.

Part 2: Phase II study to evaluate the antitumor efficacy of SY-5007. Patients with advanced RET Fusion-Positive NSCLC will be enrolled in this phase. SY-5007 will be administered orally 160mg twice daily in a 28-day cycle. This phase is designed to determine the antitumor activity (ORR, DCR, DoR, PFS and OS), safety, and PK of SY-5007.

ELIGIBILITY:
Inclusion Criteria:

-

For Phase I:

1. Male or female, at least 18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
3. Estimated life expectancy >12 weeks.
4. Patients must have at least one assessable lesion in dose-escalation part and one measurable lesion in dose-expansion part per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
5. Dose-escalation Part: patients must have histological or cytological confirmed advanced solid tumours with RET alteration (fusion or mutation) and have progressed after standard therapy, or no standard or available curative therapy exists.

   Dose-expansion Part: Patients with advanced tumor must have histological or cytological confirmed RET alteration, including NSCLC patients with RET-fusion or MTC patients with RET-mutation or other patients with RET alteration, and either have progressed after standard therapy or no standard/ available curative therapy exists.
6. Patients must have adequate organ function as defined in the below:

   Hepatic function:

   Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN) if no hepatic metastases are present, or otherwise ≤ 5 times ULN, Total serum bilirubin (TBIL) ≤ 1.5 times ULN.

   Bone marrow function (No blood transfusion or haematopoietic stimulating factor treatment within 10 days prior to testing):

   Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L; Platelets (PLT) count ≥ 75 x 10⁹/L; Hemoglobin (Hb) ≥ 85 g/L.

   Renal function:

   Creatinine clearance ≥ 50 mL/min.

   Coagulation function:

   Prothrombin time (PT) or International Normalized Ratio (INR) ≤ 1.5 times ULN.

   Serum lipid:

   Cholesterol ≤ 500mg/dL（12.92mmol/L）.
7. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to the first dose, male and female patients of childbearing potential must be willing to completely abstain or agree to use an appropriate method of contraception during the entire study duration and for at least 3 months after the last dose of study medication.
8. Willingness and ability to give informed consent and follow protocol procedures, and comply with follow-up visit requirements.

   For Phase II: As for phase I with the following modifications:
9. Participants must have histological or cytological confirmed locally advanced or metastatic RET Fusion-Positive NSCLC, have progressed following platinum-based chemotherapy and/or PD-1/PD-L1 immunotherapy, or have not received prior systemic therapy, or in the opinion of the Investigator, they would be unlikely to tolerate or derive significant clinical benefit from appropriate standard of care therapy, or they declined standard therapy.
10. The participants' tumor tissue or blood sample test results meet 1 of the following 2 criteria:

    1. Previous tumor tissue or blood sample confirmed positive for RET fusion by local laboratory.
    2. If no previous positive RET fusion test report is available, a compliant tumor tissue or blood sample must be tested at a central laboratory designated by the sponsor, using a second-generation sequencing (NGS)-based assay, and confirmed as positive for RET fusion.

Exclusion Criteria:

1. Dose-expansion Part: Patient's cancer has a known primary driver alteration other than RET. e.g. EGFR, ALK, ROS1, KRAS, etc.
2. Dose-expansion Part: Patients previously treated with a selective RET inhibitor.
3. Patients received systemic antitumor therapy, including chemotherapy, radiotherapy, biologic therapy, endocrine therapy, or immunotherapy within 3 weeks prior to the first dose, except for the following:

   Nitrosoureas or mitomycin C within 6 weeks; Oral fluorouracils and small molecule drugs within 2 weeks or within 5 half-life periods of the drug (whichever is longer); Antitumour traditional Chinese medicine within 2 weeks.
4. Patients received other unlisted clinical trial drugs or treatments within 4 weeks prior to the first dose.
5. Patients underwent major organ surgery (excluding puncture biopsy) or had significant trauma within 4 weeks prior to the first dose.
6. Adverse effects of previous anti-tumor therapy have not recovered to CTCAE 5.0 grade rating of ≤ grade 1 (except for toxicity judged by the investigator be of no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, etc.)
7. Patients have symptomatic central nervous system (CNS) metastases, meningeal metastases, or a primary CNS tumor that is associated with progressive neurological symptoms.
8. Patients with active uncontrolled systemic bacterial, viral, or fungal infection despite optimal treatment (chronic disease screening not required).
9. Active hepatitis (Hepatitis B: HBsAg-positive and HBV-DNA ≥ 2000 IU/ mL; Hepatitis B: HCV antibody-positive and HCV-RNA ≥ 1000 IU/ml), HIV antibody-positive; Active syphilis.
10. Patients have a history of severe cardiovascular disease, including but not limited to:

    Severe cardiac rhythm or conduction abnormalities, e.g. ventricular arrhythmia requiring clinical intervention, II-III degree atrioventricular block, etc.

    Mean QT interval corrected using Fridericia's formula (QTcF)> 480ms at rest. Acute coronary syndrome, congestive heart failure, aortic coarctation, stroke or other grade 3 or higher cardiovascular or cerebrovascular events within 6 months prior to the first dose.

    New York Heart Association (NYHA) ≥ class II heart failure or left ventricular ejection fraction (LVEF) < 50%.

    Hypertension remains uncontrolled after aggressive antihypertensive therapy.
11. Patients have been treated with any CYP3A inhibitors or inducers within 14 days prior to the first dose.
12. Patients with malignancies other than tumors treated in this study (except: malignancies that are cured and have not recurred within 3 years prior to study entry; completely resected basal cell and squamous cell skin cancer; completely resected carcinoma in situ of any type).
13. Patients are unable to swallow the drug orally, or has a condition that seriously affects gastrointestinal absorption in the judgment of the investigator.

    For Phase II: As for phase I with the following modifications:
14. Patients received any selective RET inhibitor (including marketed drugs such as selpercatinib, pralsetinib, and unmarketed experimental drugs).
15. Patients have a history of hypersensitivity to any component or excipient of SY-5007 capsule.
16. Patients participated in another clinical study within 4 weeks prior to the first dose or is scheduled to participate in another clinical study during the study period.
17. Pregnant or breastfeeding female patients.
18. Other conditions deemed by the investigator to be inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Phase I: Determine the dose-limiting toxicities (DLT) during the first 28-day cycle of SY-5007 treatment | Dose-escalation Cycle 1 (each cycle is 28 days)
  Maximum Tolerated Dose (MTD) and/or recommended phase 2 dose (RP2D) in Cycle 1
Phase I: Number of patients with adverse events and serious adverse events | Up to 24 months
  Characterization of the safety and tolerability
Phase II: Overall Response Rate (ORR) as assessed by RECIST 1.1 criteria | Up to 24 months
  Anti-tumor activity of SY-5007

SECONDARY OUTCOMES:
Phase I: Overall Response Rate (ORR) as assessed by RECIST 1.1 criteriaOverall Response Rate (ORR) as assessed by RECIST 1.1 criteria | Up to 24 months
  Preliminary anti-tumor activity of SY-5007
Phase I & II: Disease control rate (DCR) as assessed by RECIST 1.1 criteria | Up to 24 months
  Preliminary anti-tumor activity of SY-5007
Phase I & II: Duration of response (DOR) | Up to 24 months
  Preliminary anti-tumor activity of SY-5007
Phase I & II: Progression Free Survival (PFS) | Up to 24 months
  Preliminary anti-tumor activity of SY-5007
Phase I & II: Overall survival (OS) | Up to 24 months
  Anti-tumor activity of SY-5007
Phase I & II: Percentage of Participants with any Serious Adverse Events (SAEs) | Up to 24 months
  Characterization of the safety and tolerability
Phase I & II: Pharmacokinetic Parameters Including Maximum Plasma Drug Concentration (Cmax) | Protocol-defined time points during Cycles 1 and 2 of treatment, up to approximately 2 months per subject
  Cmax of SY-5007
Phase I & II: Pharmacokinetic Parameters Including time to maximum plasma concentration (Tmax) of SY-5007 | Protocol-defined time points during Cycles 1 and 2 of treatment, up to approximately 2 months per subject
  Tmax of SY-5007
Phase I & II: Pharmacokinetic Parameters Including Area Under the Plasma Concentration-Time Curve of SY-5007 (AUC) | Protocol-defined time points during Cycles 1 and 2 of treatment, up to approximately 2 months per subject
  AUC of SY-5007
Phase I & II: Pharmacokinetic Parameters Including Terminal Elimination Half-life (t1/2) of SY-5007 | Protocol-defined time points during Cycles 1 and 2 of treatment, up to approximately 2 months per subject
  plasma terminal phase disposition half-life of SY-5007

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, PhD, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (2):
- China (2):
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Li W, Wang Y, Xiong A, Gao G, Song Z, Zhang Y, Huang D, Ye F, Wang Q, Li Z, Liu J, Xu C, Sun Y, Liu X, Zhou F, Zhou C. First-in-human, phase 1 dose-escalation and dose-expansion study of a RET inhibitor SY-5007 in patients with advanced RET-altered solid tumors. Signal Transduct Target Ther. 2024 Nov 4;9(1):300. doi: 10.1038/s41392-024-02006-9. PMID 39489747